CLINICAL TRIAL: NCT03017066
Title: Ultrasound Assessment of Gastric Volume Following Preoperative Fasting Guideline in Pediatric Patients
Brief Title: Ultrasound Assessment of Preoperative Gastric Volume in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Associate professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1612100815
Record Dates: First submitted 2017-01-05; First posted 2017-01-11 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Fasting
Keywords: Ultrasonography; Child; Preoperative period
MeSH Terms: conditions — Fasting | interventions — Ultrasonography; Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infant formula (Experimental): Patients were given infant formula 6 hours prior to surgery. Gastric volume was assessed before ingestion, 1 hour prior to the surgery, and before the induction of general anesthesia using ultrasound.
  Interventions: Device: Ultrasound; Other: General anesthesia
- Carbohydrate drink (Experimental): Patients were given carbohydrate drink 2 hours prior to surgery. Gastric volume was assessed before ingestion, 1 hour prior to the surgery, and before the induction of general anesthesia using ultrasound.
  Interventions: Device: Ultrasound; Other: General anesthesia

INTERVENTIONS:
Device: Ultrasound — Ultrasound assessment of gastric volume is performed three times; before ingestion of infant formula or carbohydrate drink; 1 hour prior to the surgery; and before induction of general anesthesia.
Other: General anesthesia — Scheduled operation under general anesthesia

SUMMARY:
The purpose of this study is to compare the gastric volume in pediatric patients who followed preoperative fasting guideline using ultrasound.

ELIGIBILITY:
Inclusion Criteria:

- Pediatric patients scheduled for elective orthopedic, otolaryngologic, ophthalmologic, plastic, and urologic surgery under general anesthesia

Exclusion Criteria:

* History of surgery on the esophagus or stomach
* History of gastrointestinal disease
* Ambulatory surgery
* Considered inappropriate by the investigator

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-04-20 (Actual)

PRIMARY OUTCOMES:
Intra-group difference between gastric volume measured on second and third ultrasound assessment | Interval between second and third ultrasound assessment, an expected average of 1 hour

SECONDARY OUTCOMES:
Inter-group difference in gastric volume at each time point | From 6 hours prior to surgery to the induction of general anesthesia, an expected average of 6 hours
Perioperative incidence of nausea, vomiting, fever, and respiratory complications | From the induction of general anesthesia until postoperative 24 hours
Degree of patient's preoperative anxiety, scored from 0 to 10, with 0 being good and 10 being bad | From 8 hours prior to surgery to the induction of general anesthesia, an expected average of 8 hours
Degree of patient's preoperative hunger, scored from 0 to 10, with 0 being good and 10 being bad | From 8 hours prior to surgery to the induction of general anesthesia, an expected average of 8 hours
Degree of patient's preoperative nausea, scored from 0 to 10, with 0 being good and 10 being bad | From 8 hours prior to surgery to the induction of general anesthesia, an expected average of 8 hours
Degree of patient's preoperative thirst, scored from 0 to 10, with 0 being good and 10 being bad | From 8 hours prior to surgery to the induction of general anesthesia, an expected average of 8 hours
Degree of patient's preoperative weakness, scored from 0 to 10, with 0 being good and 10 being bad | From 8 hours prior to surgery to the induction of general anesthesia, an expected average of 8 hours
Degree of patient's preoperative irritability, scored from 0 to 10, with 0 being good and 10 being bad | From 8 hours prior to surgery to the induction of general anesthesia, an expected average of 8 hours
Degree of parent's satisfaction, scored from 0 to 10, with 0 being satisfied and 10 being unsatisfied | From 8 hours prior to surgery to the induction of general anesthesia, an expected average of 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perlas A, Chan VW, Lupu CM, Mitsakakis N, Hanbidge A. Ultrasound assessment of gastric content and volume. Anesthesiology. 2009 Jul;111(1):82-9. doi: 10.1097/ALN.0b013e3181a97250. PMID 19512861
- [Background] Bouvet L, Mazoit JX, Chassard D, Allaouchiche B, Boselli E, Benhamou D. Clinical assessment of the ultrasonographic measurement of antral area for estimating preoperative gastric content and volume. Anesthesiology. 2011 May;114(5):1086-92. doi: 10.1097/ALN.0b013e31820dee48. PMID 21364462
- [Background] Fukunaga C, Sugita M, Yamamoto T. Validity of ultrasonographic measurement of gastric volume in fasted pediatric patients without sedation. J Anesth. 2016 Oct;30(5):900-3. doi: 10.1007/s00540-016-2204-3. Epub 2016 Jun 22. PMID 27334390
- [Background] American Society of Anesthesiologists Committee. Practice guidelines for preoperative fasting and the use of pharmacologic agents to reduce the risk of pulmonary aspiration: application to healthy patients undergoing elective procedures: an updated report by the American Society of Anesthesiologists Committee on Standards and Practice Parameters. Anesthesiology. 2011 Mar;114(3):495-511. doi: 10.1097/ALN.0b013e3181fcbfd9. No abstract available. PMID 21307770
- [Background] Smith I, Kranke P, Murat I, Smith A, O'Sullivan G, Soreide E, Spies C, in't Veld B; European Society of Anaesthesiology. Perioperative fasting in adults and children: guidelines from the European Society of Anaesthesiology. Eur J Anaesthesiol. 2011 Aug;28(8):556-69. doi: 10.1097/EJA.0b013e3283495ba1. PMID 21712716
- [Background] Brady M, Kinn S, Ness V, O'Rourke K, Randhawa N, Stuart P. Preoperative fasting for preventing perioperative complications in children. Cochrane Database Syst Rev. 2009 Oct 7;(4):CD005285. doi: 10.1002/14651858.CD005285.pub2. PMID 19821343
- [Background] Brunet-Wood K, Simons M, Evasiuk A, Mazurak V, Dicken B, Ridley D, Larsen B. Surgical fasting guidelines in children: Are we putting them into practice? J Pediatr Surg. 2016 Aug;51(8):1298-302. doi: 10.1016/j.jpedsurg.2016.04.006. Epub 2016 Apr 21. PMID 27166876